CLINICAL TRIAL: NCT03859466
Title: Safety and Efficacy of Cardiac Shockwave Therapy in Patients Undergoing Coronary Artery Bypass Grafting
Acronym: CAST-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP-HEART-001
Record Dates: First submitted 2018-11-08; First posted 2019-03-01 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure Patients; Cardiac Ischemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: This study investigates the safety and performance characteristics of the Direct Epicardial Shockwave Therapy System (DESWT) as applied with the Cardiac Shockwave Probe (CSP) vs. Sham treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking is performed using opaque envelopes that are opened by an assistant at the end of the CABG procedure after the bypasses are fully established.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): In the intervention arm, 300 shockwave impulses per coronary supply territory, at an energy flux density of 0.38mJ/mm2 and a frequency 3Hz, are applied in direct contact with the ischaemic myocardium of the left ventricle. The intervention is performed during CABG surgery after bypasses are fully established while still on cardiopulmonary bypass.
  Interventions: Device: Shockwave Therapy
- Sham Control Arm (No Intervention): In the sham control arm, the same manipulations are performed with an inactive shockwave applicator in direct contact with the ischaemic myocardium of the left ventricle as in the intervention arm. The sham treatment is performed during CABG surgery after bypasses are fully established while still on cardiopulmonary bypass.

INTERVENTIONS:
Device: Shockwave Therapy — The cardiac shockwave system consists of a table-top device (Nonvasiv Medical GmbH, Konstanz, Germany) and a sterile single-use applicator releasing electrohydraulic shockwaves (Heart Regeneration Technologies GmbH, Innsbruck, Austria). Prior to use, the applicator is inserted into a sterile cover containing ultrasound gel. In order to ensure acoustic coupling between the applicator and the myocardium, continuous saline rinsing is applied throughout the procedure.
  Arms: Intervention Arm

SUMMARY:
This randomised, controlled clinical trial aims to evaluate the safety and efficacy of Cardiac Shockwave Therapy (CAST-HF) in patients with ischaemic heart failure requiring surgical revascularization. The main questions to answer are:

* Does cardiac shockwave therapy, in addition to CABG surgery, improve left ventricular ejection fraction?
* Is cardiac shockwave therapy in addition to CAGB surgery safe?

Participants will be randomised into intervention (cardiac shockwave therapy) and control (sham treatment with an inactive applicator) groups.

DETAILED DESCRIPTION:
This study investigates the safety and performance characteristics of the Direct Epicardial Shockwave Therapy System (DESWT) as applied with the Cardiac Shockwave Probe (CSP).

ELIGIBILITY:
Inclusion criteria

* Male or female patients between 21 and 90 years of age undergoing primary coronary artery bypass grafting
* Presentation with reduced left ventricular function, defined as LVEF ≤ 40% measured by cardiac MRI
* Presentation with regional left ventricular wall motion abnormalities
* Written informed consent from the patient for participation in the study

Exclusion criteria

* Significant concomitant aortic valve disease requiring surgical treatment (other than significant aortic valve disease not detected in preoperative cardiac ultrasound but detected during surgery)
* Serious radiographic contrast allergy
* Patient in cardiogenic shock or presenting with acute myocardial infarction (STEMI or NSTEMI)
* Patient with a contraindication for cardiac MRI
* History of significant ventricular arrhythmia, other than MI-associated arrhythmia
* Comorbidity reducing life expectancy to less than one year
* Presence of a ventricular thrombus
* Presence of a cardiac tumour
* Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the improvement in LVEF measured by cardiac MRI from baseline to 360 days. | 360 days
  The primary efficacy objective is to assess the efficacy of cardiac shock wave therapy in patients undergoing primary coronary artery bypass grafting and suffering from reduced left ventricular function ≤ 40%
The primary safety endpoint is the occurrence of device-related complications (adverse device effects or serious adverse device effects) within 360 days. | 360 days
  The primary safety objective is to assess the safety profile of the cardiac shock wave therapy device.

SECONDARY OUTCOMES:
Secondary efficacy-related endpoints include patient-reported outcomes. | 360 days
  Change in:
  * 6- Minute Walk Test Distance
  * NYHA functional class
  * Serum nt-proBNP levels
  * Renal function (GFR)
  * Seattle Angina Pectoris Questionnaire (SAQ)
  * 36-item short-form survey (SF36)
  * Minnesota Living with Heart Failure Questionnaire (MLHFQ)
Secondary safety-related endpoints include patient-reported outcomes. | 6 Days
  * Occurance of ventricular arrhythmia during hospital stay
  * Occurrence of device-related peri-operative myocardial damage detected by rise of cardiac biomarkers (CK-MB, TropT) Occurrence of signs of device-related infection (CRP, leucocytosis) during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Holfeld, MD, Principal Investigator — University Hospital for Cardiac Surgery, Medical University of Innsbruck, Innsbruck, Austria
Locations (1):
- Medical University of Innsbruck - Competence Center for Clinical Trials, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Nagele F, Polzl L, Graber M, Hirsch J, Mayr A, Pamminger M, Troger F, Theurl M, Schreinlechner M, Sappler N, Dorfmuller C, Mitrovic M, Ulmer H, Grimm M, Gollmann-Tepekoylu C, Holfeld J. Safety and efficacy of direct cardiac shockwave therapy in patients with ischemic cardiomyopathy undergoing coronary artery bypass grafting (the CAST-HF trial): study protocol for a randomized controlled trial-an update. Trials. 2022 Dec 9;23(1):988. doi: 10.1186/s13063-022-06931-4. PMID 36494706
- [Derived] Polzl L, Nagele F, Graber M, Hirsch J, Lobenwein D, Mitrovic M, Mayr A, Theurl M, Schreinlechner M, Pamminger M, Dorfmuller C, Grimm M, Gollmann-Tepekoylu C, Holfeld J. Safety and efficacy of direct Cardiac Shockwave Therapy in patients with ischemic cardiomyopathy undergoing coronary artery bypass grafting (the CAST-HF trial): study protocol for a randomized controlled trial. Trials. 2020 May 30;21(1):447. doi: 10.1186/s13063-020-04369-0. PMID 32473644
- See also: Cardiac Regeneration Research Lab — http://www.carelab.at
- See also: Trial Homepage — http://www.cast-trial.com